CLINICAL TRIAL: NCT04040218
Title: Harms Associated With Dry Needling Provided During Patient Care in Colorado by Physical Therapists
Brief Title: Trigger Point Dry Needling Practice in Colorado: Practitioner and Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regis University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 1069837-1
Record Dates: First submitted 2019-07-30; First posted 2019-07-31 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Dry Needling; Harm
Keywords: dry needling; physical therapy
MeSH Terms: interventions — Dry Needling

STUDY DESIGN:
Intervention Model Description: The target population for this study was a representative sample of PT providers that administer and patients that receive dry needling as a treatment modality in the state of Colorado. 440 PT's licensed in Colorado and 2167 patients were recruited for this study. Purposive sampling was implemented through convenience sampling methods; by which PT respondents were included through their association to APTA CO or Kinetacore@ (an education provider in DN) and patients through their PT provider. The PT survey was sent out to APTA CO members and via a Kinetacore email list; which included approximately 900 individuals trained by Kinetacore in CO. All respondents to the PT survey were requested to provide patients with a direct link to the patient survey. Invitation was promoted by APTA CO outside of their member portal to non-members and word of mouth was encouraged.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Dry Needling — Dry needling is utilized by multiple practitioners to address impairments in neuromusculoskeletal function, often related to pain and loss of mobility. Dry needling, according the American Physical Therapy Association (APTA), is defined as a skilled intervention that uses a thin filiform needle to penetrate the skin and stimulate underlying myofascial trigger points, muscular, and connective tissues for the management of neuromusculoskeletal pain and movement impairments

SUMMARY:
A retrospective analysis of responses following a descriptive survey to investigate the benefits and harms associated with dry needling as provided by a physical therapists in CO

DETAILED DESCRIPTION:
Two surveys were completed to identify the reported harms by physical therapists in the provision of dry needling in Colorado, and by patients who received dry needling from physical therapists in Colorado in April 2017. Retrospective analysis of the data (de-identified) was completed to provide a representative reporting on harms associated with the dry needling provided and received for patients.

ELIGIBILITY:
Inclusion Criteria:

* Physical therapists providing dry needling to patients in Colorado
* Patients who had received dry needling from Physical Therapists in Colorado

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2607 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
Survey analysis of harm data | As reported during the four week survey time frame
  Harm - "any ill-effect, no matter how small, that was unintended." Further delineation was made that minor/insignificant complaints/harms were defined as short term soreness less than 24 hours and more than 24 hours, bruising and light-headedness, and major/significant harm was defined infection or pneumothorax (PTX).

CONTACTS AND LOCATIONS:
Locations (1):
- Regis University, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No